CLINICAL TRIAL: NCT01658553
Title: A Phase I, Single-Sequence, Placebo-Controlled, Single-Blind Study to Evaluate the Effect of Repeat Oral Dosing of GSK1120212 on Cardiac Repolarization in Subjects With Solid Tumors
Brief Title: A Study to Look at the Electrical Activity of the Heart in Subjects With Solid Tumor Cancers, Before and After Receiving the Study Treatment, GSK1120212
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 114655
Record Dates: First submitted 2012-06-28; First posted 2012-08-07 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Cancer
Keywords: solid tumors
MeSH Terms: conditions — Neoplasms | interventions — trametinib

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK1120212 Qtc study (Experimental): Single-Sequence, Placebo-Controlled, Single-Blind Study to Evaluate the Effect of Repeat Oral Dosing of GSK1120212 on Cardiac Repolarization in Subjects with Solid Tumors
  Interventions: Drug: GSK1120212

INTERVENTIONS:
Drug: GSK1120212 — GSK1120212 - placebo match oral dose on day 1 with GSK1120212 3 mg oral dose on day 15. GSK1120212 2mg and 2 tablets of GSK1120212 -placebo matched 0.5 mg oral dose daily from day 2 to day 14. 24 hour holter monitoring will be performed on day 1 and day 15 to compare the subjects cardiac repolarization while on placebo and after having received GSK1120212 for 14 days

SUMMARY:
A multicenter, non-randomized, placebo-controlled, single dosing schedule, subject-blinded study to evaluate the effect of GSK1120212 on the electrical activity of the heart as compared to placebo in subjects with solid tumor cancers. All subjects will undergo Screening assessments within 21 days prior to the start of the study treatment to determine their eligibility for enrollment in the study. Eligible subjects will receive study treatment administered over a period of 15 days followed by a post-treatment follow-up visit. Study treatment (GSK1120212-matched placebo) will be blinded to subjects. Subjects will receive GSK1120212-matched placebo on one day during the first 14 days of dosing. On all other days the subject will receive a once-daily 2 mg dose of GSK1120212 except for Day 15 when the subject will receive 3mg dose of GSK1120212 12-lead ECG recordings will be obtained from continuous ECG recordings obtained via a 12-lead Holter monitor on Study Days 1 and 15 while subjects are in the clinical research unit. The effect of GSK1120212 on the electrical activity of the heart will be determined by time-matched ECGs obtained at the same time points relative to dosing on these days. Ambulatory blood pressure readings will be obtained from continuous 24-hour recordings via an ambulatory blood pressure monitor The effect of GSK1120212 on blood pressure parameters will be determined by blood pressure readings obtained at the same time points relative to dosing on Study Days 1 and 15. Serial blood samples to analyze the concentration of study drug in the subject's blood will be obtained at the same time points relative to dosing on Study Days 1 and 15. Subjects who are eligible for continued treatment with GSK1120212 may continue treatment under the rollover study MEK114375 (drug study number). A post-treatment follow-up visit will be conducted within 28 days of the last dose of study treatment for all subjects who do not continue treatment in the rollover study MEK114375.

DETAILED DESCRIPTION:
GSK1120212 is an orally administered, potent and highly selective small molecule inhibitor of MEK1(mitogen-activated extracellular signal-regulated kinase-1)/MEK2 (mitogen-activated extracellular signal-regulated kinase-2) activation and kinase activity. As monotherapy, GSK1120212 has shown an acceptable risk-benefit profile with encouraging efficacy in various oncologic settings. This Phase I, single-sequence, placebo-controlled, singleblind, multicenter study is designed to evaluate the effects of repeat oral dosing of GSK1120212 on electrocardiographic parameters with a particular focus on its effect on cardiac repolarization (Corrected QT interval [QTc] duration) as compared to placebo in subjects with solid tumor cancers. A single dose of placebo will be administered on Study Day 1 followed by administration of a once-daily 2 mg dose of GSK1120212 for 13 days (Study Days 2 through 14) and on Study Day 15 a dose of 3 mg of GSK1120212 will be given. Digital 12-lead electrocardiograms (ECGs) will be extracted from continuous ECG recordings obtained via Holter monitor on Study Days 1 and 2 after the administration of placebo and on Study Days 15 and 16 after the administration of GSK1120212. Pharmacokinetic samples will be time-matched with the Holter ECGs. This study will also assess the exposure-QTc relationship between plasma concentrations of GSK1120212 and its effect, if any, on cardiac repolarization, specifically on the QTc interval. Continuous 24-hour ambulatory blood pressure monitoring will be conducted to assess the effect of GSK1120212 on blood pressure parameters on Study Days 1 and 15. Safety assessments, including assessment of adverse events, clinical laboratory tests (hematology and clinical chemistry) and vital signs, will be performed throughout the study. Following completion of study treatment, eligible subjects may transition to the open-label, rollover study MEK114375 to continue treatment with GSK1120212.

ELIGIBILITY:
Inclusion Criteria

* Has provided signed, written informed consent.
* Male or female, age greater than and equal to 18 years of age at the time of signing the informed consent form.
* Has histologically or cytologically confirmed diagnosis of a solid tumor malignancy that is not responsive to standard therapy(ies) or for which there is no approved therapy.
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Able to swallow and retain oral medication.
* Has adequate baseline organ function as follows: System: Hematologic - absolute neutrophil count, Laboratory values: greater than and equal to 1.2 × 109/L;System: Hematologic - Hemoglobin, laboratory values: greater than and equal to 9 g/dL; System: Hematologic-platelets, laboratory values: greater than and equal to 75 × 109/L; System: Hematologic - Prothrombin time (PT), INR (international normalizing ratio - a blood clotting test))and Partial thromboplastin time (PTT), laboratory values: less than and equal to 1.5 times ULN(Upper limit of normal); System - Hepatic - Total bilirubin, laboratory values: less than and equal to 1.5 times ULN; System: Hepatic-ALT(Alanine aminotransferase), laboratory values: less than and equal to 2.5 times ULN; System: Renal-Creatine, laboratory values: less than anad equal to 1.5 times ULN; or System: Renal-Calculated creatinine clearance, laboratory values: greater than and equal to 50 mL/min; or System: Renal-24hour urine creatine clearance, laboratory values: greater than and equal to 50 mL/min; System: Cardiac-LVEF, laboratory values: greater than and equal to LLN (Lower limit of normal) by ECHO or MUGA(Multigated acquisition scan). Abbreviations: ALT, alanine aminotransferase; AST, aspartate aminotransferase; ECHO, echocardiogram; INR; LLN,lower limit of normal; LVEF, left ventricular ejection fraction; MUGA; PT, prothrombin time; PTT, partial thromboplastin time; ULN, upper limit of normal. INR greater than 1.5 times ULN will be acceptable in case of subjects receiving therapeutic anticoagulants such as warfarin as long as INR is monitored during the study according to clinical practice; Calculated by the Cockcroft-Gault formula; If LLN is not defined for a given institution, then ejection fraction must be greater than and equal to 50%. NOTE: Subjects with aspartate aminotransferase (AST), ALT or bilirubin values outside the range(s) in the table due to Gilbert's syndrome or asymptomatic gallstones are not excluded. Laboratory results obtained during Screening should be used to determine eligibility criteria. In situations where laboratory results are outside the permitted range, the investigator may opt to retest the subject and the subsequent within-range screening result may be used to confirm eligibility.
* Have serum potassium, serum magnesium, and total serum calcium levels within normal limits. NOTE: If total serum calcium is below the LLN, then it will be necessary to determine the albumin-corrected total serum calcium level. Use the following calculation: Calcium (mg/dL) = measured total Calcium (mg/dL) + 0.8 (4.0 - serum albumin [g/dL]) NOTE: If serum potassium or magnesium level is below the LLN, supplementation is permitted in order to meet the inclusion criterion. Subject should be retested following supplementation. In order to avoid a situation where the subject cannot be dosed during the study due to electrolyte levels falling below the LLN, it is strongly recommended to maintain serum potassium levels greater than 4 mEq(Milliequivalent )/L and serum magnesium levels greater than 2.2 mg/dL whenever possible. Slight elevations of potassium or magnesium above the upper limit of normal may be seen during supplementation and will not exclude subjects from study entry.
* If a female subject of childbearing potential, must have a negative serum pregnancy test within 14 days of first dose of study treatment and agree to use effective contraception, as defined in the protocol. during the study and for 4 months following the last dose of study treatment.

Exclusion Criteria:

* History of prior exposure to a MEK(activated extracellular signal-regulated kinase) inhibitor or disease progression while receiving treatment with a MEK inhibitor.
* Any of the following ECG findings: QTcF (preferred) or QTcB(interval corrected for heart rate by Bazett's formula) interval greater than and equal to 480 msec; PR(Partial response) interval greater than 220 msec or less than and equal to 110 msec; Bradycardia defined as sinus rate less than 50 beats per minute (bpm)
* Cardiac conduction abnormalities denoted by any of the following: Evidence of second-degree (type II) or third-degree atrioventricular block; Evidence of ventricular pre-excitation; Electrocardiographic evidence of complete left bundle branch block (LBBB) NOTE: Right bundle branch block (RBBB), incomplete LBBB or incomplete RBBB will be exclusionary ONLY if QRS(a name for the combination of the graphical deflections seen on a typical electrocardiogram) duration is greater than 120 msec; Intraventricular conduction delay with QRS duration greater than 120 msec; Evidence of atrial fibrillation or history of atrial fibrillation within the past 6 months; Presence of cardiac pacemaker
* History or evidence of any one of the following cardiovascular conditions within the past 6 months: Class II, III, IV heart failure as defined by the New York Heart Association; Cardiac angioplasty or stenting; Myocardial infarction; Unstable angina; Symptomatic peripheral vascular disease or other clinically significant cardiac disease; Cardiac metastases
* Left ventricular ejection fraction (LVEF), as measured by ECHO or MUGA scan, below the institutional LLN, or if a LLN does not exist at an institution, less than 50%
* Personal or family history of long-QT syndrome.
* Treatment-refractory hypertension defined as a blood pressure of SBP (Systolic blood pressure) greater than 140 mmHg and/or DBP(Diastolic blood pressure) greater than 90 mmHg which cannot be controlled by anti-hypertensive therapy or lifestyle modifications.
* Anti-cancer therapy (e.g., chemotherapy with delayed toxicity, extensive radiation therapy, immunotherapy, biologic therapy, or major surgery) within 21 days prior to enrollment; chemotherapy regimens without delayed toxicity within 14 days prior to enrollment; or use of an investigational anti-cancer drug within 28 days preceding the first dose of study treatment. NOTE: Subjects with a history of prior anthracycline exposure are excluded.
* Current use of a prohibited medication(s) or requires any of these medications during treatment with study treatment. NOTE: This includes medications that are listed as drugs that are generally accepted by the QTdrug.org (Advisory Board of the Arizona Center for Education and Research on Therapeutics to have a risk of causing Torsade de pointes (available at: http://www.azcert.org/medical-pros/drug-lists/bycategory.cfm).
* Current use of therapeutic warfarin. NOTE: Low molecular weight heparin and prophylactic low-dose warfarin are permitted.
* Any unresolved toxicity of greater than and equal to Grade 2, except alopecia or Grade 2 anemia, (NCI-CTCAE), version 4.0, from previous anti-cancer therapy.
* Pre-existing Grade 2 or greater peripheral neuropathy.
* History or current evidence/risk of RVO or CSR: History of RVO (Retinal vein occlusion) or CSR (Central serous retinopathy), or predisposing factors to RVO or CSR (i.e., uncontrolled glaucoma or ocular hypertension, uncontrolled systemic disease such as hypertension or diabetes mellitus, or history of hyperviscosity or hypercoagulability syndromes); Visible retinal pathology as assessed by ophthalmic examination that is considered a risk factor for RVO or CSR such as: Evidence of new optic disc cupping; Intraocular pressure >21 mmHg as measured by tonography
* History of interstitial lung disease or pneumonitis.
* Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression. NOTE: Subjects previously treated for these conditions that have had stable central nervous system disease (verified with consecutive imaging studies) for greater than 3 months, are asymptomatic and are not currently taking corticosteroids, or are on stable dose of corticosteroids for at least 30 days prior to Study Day 1 are permitted.
* Presence of clinically significant gastrointestinal (GI) abnormalities that may affect the absorption of study treatment(s) including, but not limited to: Active, uncontrolled GI disease; Malabsorption syndrome; Substantial resection of the stomach, small bowel or colon. If clarification is needed as to whether a condition will significantly affect the absorption of study treatment(s), contact the GSK Medical Monitor.
* History or presence of hepatic insufficiency (excluding metastatic hepatic carcinoma).
* Uncontrolled medical conditions (i.e., diabetes mellitus, hypertension), psychological,familial, sociological, or geographical conditions that do not permit compliance with the protocol; or unwillingness or inability to follow the procedures required in the protocol.
* Lactating or actively breastfeeding females.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to DMSO (Dimethyl Sulfoxide).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-09-19 (Actual); Primary Completion 2014-04-05 (Actual); Study Completion 2014-04-05 (Actual)

PRIMARY OUTCOMES:
Compare the effect of GSK1120212 on the baseline-adjusted, placebo-corrected, time-matched QTcF(QT interval corrected for heart rate by Fridericia's formula) interval duration in subjects with solid tumor cancers | from baseline to day 15

SECONDARY OUTCOMES:
Evidence of the relationships between the change in QTc(Corrected QT interval) from baseline and the plasma concentrations of GSK1120212 and predicted change in QTc(Corrected QT interval) | From baseline as compared to study day 15
Plasma concentrations and PK (Pharmacokinetic) parameters of GSK1120212, including AUC(Area under concentration-time curve)(0-24), concentration at time t (Ct), Cmax (Maximum observed concentration) and time to Cmax (tmax). | From placebo dosing on day 1 to day 15
Safety parameters: AEs, vital sign (blood pressure, pulse rate and temperature), ECGs, and clinical laboratory assessments | From baseline until follow up(maximum 42 days)
Change in blood pressure parameters, including PP(Pulse pressure) and MABP(Mean arterial blood pressure) | from baseline to Study Day 15.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah

REFERENCES:
- See also: Results for study 114655 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114655?search=study&search_terms=114655#rs